## The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title : | Reporting and Analysis Plan for 205037: A single-centre, randomized, double-blind, dose-ascending, placebocontrolled study to evaluate the safety, tolerability, and pharmacokinetics of oral TID doses (one day) of GSK2982772 in Japanese healthy male subjects |
|---|---|
| Compound Number : | GSK2982772 |
| Effective Date : | 11-JUL-2018 |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 205037.
- This RAP is intended to describe the final analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

## RAP Author(s):

| Approver | Date | Approval Method |
|---|---|---|
| PPD | | |
| Biostatistics Group 2, Biomedical Data Sciences Japan | NA | NA |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Lead Programmer; Statistical Programming & Reporting Group, Biomedical Data Sciences Japan | 10-JUL-2018 | Pharma TMF |
| Clinical Investigation Leader/Operational Science Lead; Clinical Pharmacology Office | 09-JUL-2018 | Pharma TMF |
| Data Quality Lead; Data Practice Group,<br>Biomedical Data Sciences Japan | 10-JUL-2018 | Pharma TMF |
| PK Analyst; Clinical Pharmacology Office | 09-JUL-2018 | Pharma TMF |

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Lead Authors Line Manager; Biostatistics Group 2, Biomedical Data Sciences Japan | 11-JUL-2018 | Pharma TMF |
| Lead Programmers Line Manager; Statistical Programming & Reporting Group, Biomedical Data Sciences Japan | 11-JUL-2018 | Pharma TMF |

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | ODUCTIO | N | 5 |
| 2. | CLIMA | MADV OF | KEY PROTOCOL INFORMATION | 5 |
| ۷. | 2.1. | | s to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | | bjective(s) and Endpoint(s) | |
| | 2.3. | | esign | |
| | 2.4. | | al Hypotheses / Statistical Analyses | |
| 3. | PI AN | NFD ANA | ALYSES | 8 |
| • | 3.1. | | Analyses | |
| | 3.2. | | alyses | |
| 4. | ANAL | YSIS POI | PULATIONS | 8 |
| | 4.1. | | l Deviations | |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | | S | |
| | 5.1. | | reatment & Sub-group Display Descriptors | |
| | 5.2. | | e Definitions | |
| | 5.3. | | ation of Covariates, Other Strata and Subgroups | |
| | | 5.3.1. | Covariates and Other Strata | 10 |
| | 5.4. | | onsiderations for Data Analyses and Data Handling tions | 11 |
| 6. | CTUD | | _ATION ANALYSES | |
| Ο. | 6.1. | | | |
| | 0.1. | | w of Planned Study Population Analyses | |
| | | 6.1.1. | Details of Planned Study Population Summaries | 13 |
| 7. | | | YSES | |
| | 7.1. | Adverse | Events Analyses | |
| | | 7.1.1. | Details of Planned Adverse Events Summaries | 15 |
| | 7.2. | Clinical | Laboratory Analyses | |
| | | 7.2.1. | Details of Planned Clinical Laboratory Displays | 17 |
| | 7.3. | Other Sa | afety Analyses | 18 |
| | | 7.3.1. | Details of Planned Other Safety Displays | 18 |
| 8. | PHAR | RMACOKI | NETIC ANALYSES | 20 |
| | 8.1. | Pharma | cokinetic Analyses | 20 |
| | | 8.1.1. | Endpoint / Variables | 20 |
| | | | 8.1.1.1. Drug Concentration Measures | 20 |
| | | | 8.1.1.2. Derived Pharmacokinetic Parameters | 20 |
| | | 8.1.2. | Summary Measure | |
| | | 8.1.3. | Population of Interest | 21 |
| | | 8.1.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 8.1.5. | Statistical Analyses / Methods | 21 |
| | | | 8.1.5.1. Statistical Methodology Specification | |
| | | 8.1.6. | Details of Planned Pharmacokinetic Displays | 23 |

| 9. | APPE | NDICES | 24 |
|---|---|---|---|
| | 9.1. | Appendix 1: Protocol Deviation Management and Definitions for Per | |
| | | Protocol Population | 24 |
| | 9.2. | Appendix 2: Schedule of Activities | 25 |
| | | 9.2.1. Protocol Defined Schedule of Events | 25 |
| | 9.3. | Appendix 3: Study Phases and Treatment Emergent Adverse | |
| | | Events | |
| | | 9.3.1. Study Phases | |
| | | 9.3.1.1. Study Phases for Adverse Events | 28 |
| | | 9.3.1.2. Study Phases for Concomitant Medication | 29 |
| | 9.4. | Appendix 4: Data Display Standards & Handling Conventions | 30 |
| | | 9.4.1. Reporting Process | 30 |
| | | 9.4.2. Reporting Standards | |
| | | 9.4.3. Reporting Standards for Pharmacokinetic | |
| | 9.5. | Appendix 5: Derived and Transformed Data | 32 |
| | | 9.5.1. General | 32 |
| | | 9.5.2. Study Population | 32 |
| | | 9.5.3. Safety | |
| | 9.6. | Appendix 6: Reporting Standards for Missing Data | 34 |
| | | 9.6.1. Premature Withdrawals | 34 |
| | | 9.6.2. Handling of Missing Data | |
| | | 9.6.2.1. Handling of Missing and Partial Dates | 34 |
| | 9.7. | Appendix 7: Values of Potential Clinical Importance | 36 |
| | | 9.7.1. Laboratory Values | 36 |
| | | 9.7.2. ECG | 37 |
| | | 9.7.3. Vital Signs | |
| | 9.8. | Appendix 8: Abbreviations & Trade Marks | 38 |
| | | 9.8.1. Abbreviations | 38 |
| | | 9.8.2. Trademarks | 38 |
| | 9.9. | Appendix 9: List of Data Displays | 39 |
| | | 9.9.1. Data Display Numbering | 39 |
| | | 9.9.2. Mock Example Shell Referencing | 39 |
| | | 9.9.3. Deliverables | 39 |
| | | 9.9.4. Study Population Tables | 40 |
| | | 9.9.5. Safety Tables | 41 |
| | | 9.9.6. Pharmacokinetic Tables | |
| | | 9.9.7. Pharmacokinetic Figures | |
| | | 9.9.8. ICH Listings | |
| | 9.10. | Appendix 10: Example Mock Shells for Data Displays | |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol: 205037

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 07/JUN/2018).

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| To assess the safety and tolerability of<br>TID doses for one day of<br>GSK2982772 in Japanese healthy<br>male subjects. | <ul> <li>Adverse events (AEs)</li> <li>Change in laboratory values (clinical chemistry, haematology and urinalysis), 12-lead ECG, vital signs (blood pressure, pulse rate, and body temperature)</li> <li>Physical examinations, in including neurological examinations.</li> </ul> |
| To characterise the PK profile of TID doses for one day of GSK2982772 in Japanese healthy male subjects. | Derived PK parameters for GSK2982772, including area under the plasma drug concentration versus time curve over 24 hr (AUC(0-24)) and AUC over each dose interval (i.e. AUC(0-7), AUC(7-14) and AUC(14-24)). Maximum observed plasma drug concentration (Cmax) following each dose, time to maximum observed plasma drug concentration (Tmax) following each dose, terminal half-life (t1/2) following the third dose, observed trough plasma drug concentrations (C0, C7, C14 and C24), where data allow |

## 2.3. Study Design

| Overview | Overview of Study Design and Key Features | | | | |
|---|---|---|---|---|---|
| Group | N | Period 1 | Period 2 | Period 3 | Period 4 |
| Α | 3 | Placebo, TID | 60 mg, TID | 120 mg, TID | 240 mg, TID |
| В | 3 | 60 mg, TID | Placebo, TID | 120 mg, TID | 240 mg, TID |
| С | 3 | 60 mg, TID | 120 mg, TID | Placebo, TID | 240 mg, TID |
| D | 3 | 60 mg, TID | 120 mg, TID | 240 mg, TID | Placebo, TID |
| Scr | eening | Within 30 days pri | or to the first dosing. | | |
| | ent Period | The study will be of with subjects in-hot each treatment per and will be discha | The study will be comprised of four study periods each at least 7 days in duration with subjects in-house for 4 nights (through 72 hours after the 1st dose). During each treatment period, subjects will be admitted to the unit the day before dosing and will be discharged after completion of the 72-hour post-dose assessments. Each subject will receive oral TID doses of GSK2982772 in fasted condition in | | |
| | | each treatment pe | | GSK2982772 or plac | |
| Washo | out Period | | | ent period doses for a | n individual subject. |
| | | | | days after last study | |
| FOI | low-up | administration. If v | varranted, additional f | follow-up visits may b | e scheduled. |
| Design | | • | - | ect to subjects, invest | • |
| Features | | | | narmacist), a three tin | |
| Dosing Time & | ascending dose, randomized, placebo-controlled, 4-way crossover study. | | | | n dose is 720 mg/day<br>proposed Ph2b study.<br>he study. The doses in<br>I such that for each<br>atment (one subject<br>placebo). Assuming 2<br>Es, clinical labs, vital<br>and GSK Medical<br>Day 1, the remaining |
| Events | | | Schedule of Activities | | |
| <ul> <li>On Day 1, participants will be assigned a unique number (randomization number ascending numerical order. The randomization number encodes the participar assignment to one of the 4 groups, according to the randomization schedule generated prior to the study by the Biomedical Data Sciences Department at C Each participant will be dispensed blinded study treatment, labelled with his un randomization number, throughout the study.</li> <li>Subjects will be randomized to one of four sequences (A, B, C, and D), where treatments in the sequences are:</li> </ul> | | | s the participant's ion schedule repartment at GSK. | | |

| Overview of | Overview of Study Design and Key Features |
|---|---|
| | ○ A: Placebo TID / 60 mg TID / 120 mg TID / 240 mg TID |
| | o B: 60 mg TID / Placebo TID / 120 mg TID / 240 mg TID |
| | ○ C: 60 mg TID / 120 mg TID / Placebo TID / 240 mg TID |
| | o D: 60 mg TID / 120 mg TID / 240 mg TID / Placebo TID |
| | 0 |
| Interim | No interim analysis is planned. |
| Analysis | |

## 2.4. Statistical Hypotheses / Statistical Analyses

The objectives of this study are to evaluate safety, tolerability and pharmacokinetics of GSK2982772 in healthy Japanese subjects. No formal statistical hypotheses will be tested. Descriptive statistics will be used to assess safety and tolerability. An estimation approach will be used to address the pharmacokinetic study objectives, where point estimates and corresponding confidence intervals will be constructed.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

A review of safety data will be conducted at the end of each period.

The decision to proceed to higher dose strengths will be made by principal investigator and GSK's Medical Monitor based on assessment of safety and tolerability at the preceding dose. This review can include individual subject data.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All subjects who have a screening visit will be included | <ul> <li>Study Population</li> </ul> |
| Enrolled | <ul> <li>All subjects who passed screening and enter the study will be included.</li> <li>Note screening failures (who never passed screening even if rescreened) and subjects screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled poputation as they did not enter the study.</li> </ul> | Study Population |
| Safety | All subjects who have received at least one dose of study treatment will be included. | <ul><li>Study Population</li><li>Safety</li></ul> |
| Pharmacokinetic<br>(PK) | All subjects in the Safety population for whom a pharmacokinetic sample has been obtained and analyzed will be included. | • PK |

Refer to Appendix 9: List of Data Displays which details the population used for each display.

## 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | [RandAll NG] Data Displays for Reporting | | |
| Code Description | | Description | Order in TLF |
| A1 | GSK2982772 60 mg | GSK2982772 60 mg | 2 |
| A2 | GSK2982772 120 mg | GSK2982772 120 mg | 3 |
| A3 | GSK2982772 240 mg | GSK2982772 240 mg | 4 |
| Р | Placebo | Placebo | 1 |

#### 5.2. Baseline Definitions

Baseline definitions are applied to each period.

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

## 5.3. Examination of Covariates, Other Strata and Subgroups

#### 5.3.1. Covariates and Other Strata

The list of covariates may be used in descriptive summaries and statistical analyses. Additional covariates may also be considered.

| Category | Details |
|---|---|
| Covariates | See Section 8.1.5.1, describing pharmacokinetic analyses using statistical model |

# 5.4. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 9.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| 9.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 9.5 | Appendix 5: Derived and Transformed Data |
| 9.6 | Appendix 6: Reporting Standards for Missing Data |
| 9.7 | Appendix 7: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Enrolled or Safety population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 9: List of Data Displays.

| Display Type | Data | Displays Gene | erated |
|---|---|---|---|
| | Table | Figure | Listing |
| Subject Disposition | | | |
| Subject Disposition for the Subject Conclusion Record | Y | | Υ |
| Screening Status and Reasons for Screen Failure | Y | | Υ |
| Number of Subjects Enrolled by Country and Site ID | Y | | |
| Subjects for Whom the Treatment Blind was Broken | | | Υ |
| Planned and Actual Treatments | | | Υ |
| Protocol Deviations | | • | |
| Important Protocol Deviations | Y | | Υ |
| Inclusion/Exclusion Criteria Deviations | | | Υ |
| Population Analysed | | • | |
| Subjects Excluded from PK Population | | | Υ |
| Demographic and Baseline Characteristics | | | |
| Demographic Characteristics | Y | | Υ |
| Race and Racial Combinations | Y | | Υ |
| Age Ranges | Y | | |
| Medical Conditions and Concomitant Medications | | • | |
| Medical Conditions | | | Υ |
| Concomitant Medications | | | Υ |
| Exposure and Treatment Compliance | 1 | L | 1 |
| Exposure to Study Treatment | | | Y |
| NOTES | L | l . | L |

#### NOTES:

• Y = Yes display generated.

## 6.1.1. Details of Planned Study Population Summaries

#### **Subject Disposition**

## Subject Disposition for the Subject Conclusion Record

The number and percentage of subjects who completed the study as well as subjects who withdrew from the study will be summarized. Reason for withdrawal will also be summarized for subjects who withdrew from the study. Only the total column will appear.

## Screening Status and Reasons for Screen Failure

This will be based on Enrolled population. The number and percentage of subjects who passed screening and who failed screening and therefore were not entered into the study will be summarized along with the reasons for failure will be summarized for those subjects who failed screening. Only the total column will appear.

#### Number of Subjects Enrolled by Country and Site ID

This will be based on Enrolled population. The number of subjects summarized by Country, Site ID and Investigator name will be presented. Only the total column will appear.

#### **Protocol Deviations**

#### Important Protocol Deviations

The number and percentage of subjects who had important protocol deviations defined as part of the protocol deviation management plan for the study, will be summarized. Only the total column will appear.

#### **Demographic and Baseline Characteristics**

#### Demographic Characteristics

The number and percentage of subjects or summary statistics will be provided for each demographic characteristic and only the total column will appear: Sex, Age (years), Age Group (years), Ethnicity, Race detail, Height, Weight, and Body Mass Index. Age Group (years) will be categorized into three ('≤18', '19-64', '≥65'). Each demographic characteristic will be summarized using the minimum set of summary statistics.

#### Race and Racial Combinations

The five-high level FDA race categories and designated Asian subcategories will be summarized along with all combinations of high level categories which exist in the data. Only the total column will appear.

## Age Ranges

The number and percentage of subjects within each age range category will be provided. Only the total column will appear. Age range will be categorized into: 18-64 years, ≥65-84 years. This is based on the standard of EMA clinical trial results disclosure requirements.

## 7. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

## 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 9: List of Data Displays.

| Display Type | | Absolute | |
|---|---|---|---|
| | Sum | mary | Individual |
| | Т | F | L |
| Adverse Events (AEs) | | | |
| All AEs by SOC and PT | Y | | Y |
| All AEs by Maximum Intensity | Y | | |
| Drug-Related AEs by SOC and PT | Y | | |
| Drug-Related AEs by Maximum Intensity | Y | | |
| Subject Numbers for Individual AEs | | | Y |
| Relationship Between AE SOCs, PT and Verbatim Text | | | Y |
| Serious and Other Significant AEs | | | |
| Serious AEs | | | Y |
| AEs Leading to Withdrawal from Study | | | Y |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 7.1.1. Details of Planned Adverse Events Summaries

#### Adverse Events (AEs)

#### All AEs by SOC and PT

The number and percentage of subjects with all relevant adverse events will be summarized by MedDRA System Organ Class and Preferred Term by treatment group. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

## All AEs by Maximum Intensity by SOC and PT

The number and percentage of subjects with adverse events by intensity (e.g., mild, moderate, severe) will be summarized by MedDRA System Organ Class and Preferred Term by treatment group. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

#### Drug-related AEs by SOC and PT

The number and percentage of subjects with all drug-related adverse events will be summarized by MedDRA System Organ Class and Preferred Term. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

#### Drug-related AEs by Maximum Intensity by SOC and PT

The number and percentage of subjects with drug-related adverse events by intensity (e.g., mild, moderate, severe) will be summarized by MedDRA System Organ Class and Preferred Term. The counting of events and the percentages will be based on the number of subjects on each treatment, so subjects may appear in more than one treatment category.

## 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 9: List of Data Displays.

| Display Type | | Absolute | 9 |
|---|---|---|---|
| | Sumi | mary | Individual |
| | T | F | L |
| Chemistry | | | |
| Chemistry Changes from Baseline | Υ | | |
| Chemistry Values | Υ | | Y |
| Chemistry Data Shifts from Baseline Relative to Normal Range | Υ | | |
| All Chemistry Data for Subjects with any Value of PCI | | | Y |
| Chemistry Values of PCI | | | Υ |
| Haematology | | | |
| Haematology Changes from Baseline | Υ | | |
| Haematology Values | Υ | | Υ |
| Haematology Data Shifts from Baseline Relative to PCI Criteria | Υ | | |
| All Haematology Data for Subjects with any Value of PCI | | | Y |
| Haematology Values of PCI | | | Υ |
| Urinalysis | | | |
| Urinalysis Concentration Changes from Baseline (Gravity and pH) | Υ | | |
| Urinalysis Data (Gravity and pH) | Υ | | Y |
| Urinalysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, and Urobilinogen) | Y | | Y |
| Hepatobiliary (Liver) | | | |
| Liver Monitoring/Stopping Event Reporting | | | Y |
| Medical Conditions for Subjects with Liver Stopping Events | | | Y |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, SOC = System Organ Class, PT = Preferred
   Term
- Summary = Represents TF related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 7.2.1. Details of Planned Clinical Laboratory Displays

#### **Chemistry/Haematology Laboratory Tests**

### Laboratory Changes from Baseline and Values

Each quantitative laboratory test and the changes in value from baseline will be summarized at every assessed time point using n, mean, standard deviation, median, minimum, and maximum by treatment group.

#### Laboratory Data Shifts from Baseline Relative to PCI Criteria

The number and percentage of subjects with laboratory results within each PCI criteria category (Low, W/in Range, High) during each planned time assessment will be summarized by treatment group relative to their baseline category by laboratory test, where PCI criteria are available. The percentages are based on the number of subjects in the treatment group with data for the laboratory test at the specified planned time (n). The worst case post-baseline is used to summarize the subjects' overall worst case shifts during the post-baseline period.

## **Urinalysis Laboratory Tests**

#### *Urinalysis Concentration Changes from Baseline (Gravity and pH)*

Gravity and pH test and the changes in value from baseline will be summarized at every assessed time point using n, mean, standard deviation, median, minimum, and maximum by treatment group.

#### *Urinalysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, and Urobilinogen)*

The number and percentage of subjects with the above urinalysis results (character results) will be summarized by treatment group.

## 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 9: List of Data Displays.

| Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Summary | | Individual |
| | Т | F | L | Т | F | L |
| Neurological Examination | | | | | | |
| Neurological Examination Findings | Υ | | Υ | | | |
| ECG | | | | | | |
| ECG Findings | Υ | | Υ | | | |
| ECG Values | Υ | | Y | Υ | | |
| All ECG Values for Subjects with any Value of PCI | | | Y | | | |
| Cardiac Telemetry | Υ | | | | | |
| Cardiac Telemetry Abnormalities | Υ | | | | | |
| Clinically Significant Cardiac Telemetry Abnormalities | | | Y | | | |
| Vital Signs | | | | | | |
| Vitals Values | Υ | | Υ | Υ | | |
| All Vital Signs for Subjects with any Value of PCI | | | Υ | | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated, PCI = Potential Clinical Importance
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 7.3.1. Details of Planned Other Safety Displays

#### **ECG**

#### ECG Findings

The number and percentage of subjects with ECG findings (ECG interpretation) will be summarized by treatment group..

#### ECG Values

Each ECG parameter value and the change from baseline will be summarized by treatment group at every assessed time point using n, mean, standard deviation, median, minimum, and maximum.

#### Cardiac Telemetry

The number and percentage of subjects with telemetry result of "normal," "abnormal but clinically insignificant," and "abnormal and clinically significant" will be summarized by

treatment group. The number and percentage of subjects with specific telemetry abnormalities will be summarized by treatment group.

## **Vital Signs**

## Vital Signs

Each vital sign parameter and the changes in value from baseline will be summarized by treatment group at every assessed time point using n, mean, standard deviation, median, minimum, and maximum.

## 8. PHARMACOKINETIC ANALYSES

## 8.1. Pharmacokinetic Analyses

## 8.1.1. Endpoint / Variables

## 8.1.1.1. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 9.4.3 Reporting Standards for Pharmacokinetic)

#### 8.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin 6.3 or hihger. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| Parameter AUC(0-7), AUC(7-14), AUC(14-24), AUC(0-24) | The area under the concentration-time curve will be calculated to some fixed nominal time x (AUC(0-x), using the combination of linear and logarithmic trapezoidal methods (i.e., Linear Up/Log Down calculation method in Phoenix WinNonlin Professional). If a sampling time deviation occurred at nominal time x (and x < t), AUC(0-x) will be calculated using the concentration at time x post-dose estimated by the method of interpolation. If nominal time x > t (or if the concentration at time x was below the limit of quantification), then the concentration (y) at time x is estimated using lambda_z and last observed Ct according to the formula: y = Ct(obser) x e-lambda_z(x-t) Then the following equation will be used to calculate (AUC(0-x)) where t is the time of last quantifiable plasma concentration. AUC(0-x) = AUC(0-t) x AUC(t-x) If lambda_z is not estimable, a partial AUC is not calculated (when x > t). |
| Cmax | Maximum observed plasma concentration following each dose will be obtained directly from the concentration-time data. |
| Tmax | The time to maximum observed plasma drug concentration following each dose will be obtained directly from the concentration-time data. |
| t1/2 | Terminal half-life following the 3rd dose will be calculated as follows:<br>t1/2 = ln2 / lambda_z |
| C0 | The plasma drug concentration at 0 hour will be obtained directly from the observed concentration-time data. |
| C7 | The plasma drug concentration at 7 hours will be obtained directly from the observed concentration-time data. |
| C14 | The plasma drug concentration at 14 hours will be obtained directly from the observed concentration-time data. |
| C24 | The plasma drug concentration at 24 hours will be obtained directly from the observed concentration-time data. |

| Parameter | Parameter Description |
|---|---|
| lambda_z | The first order rate constant associated with the terminal (log-linear) portion of the curve following the 3rd dose. |
| lambda_z<br>lower | The lower limit on time for values to be included in the calculation of lambda_z following the 3rd dose |
| lambda_z<br>upper | The upper limit on time for values to be included in the calculation of lambda_z following the 3rd dose |
| #pts | The number of time points used in computing lambda_z following the 3rd dose |
| R-square | Square of the correlation coefficient for computing lambda_z following the 3rd dose. |

#### NOTES:

- Additional parameters may be included as required.
- Lambda\_z is the terminal phase rate constant.
- Ct is the last observed quantifiable concentration.

## 8.1.2. Summary Measure

The slope of log-transformed dose in the power model for AUC(0-24), AUC(0-7) and Cmax will be used as measure of the dose proportionality between dose and the PK parameters..

### 8.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

## 8.1.4. Strategy for Intercurrent (Post-Randomization) Events

Intercurrent events which may affect the assessment of the safety and tolerability and the characterization of PK profile will not be anticipated.

### 8.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 8.1.5.1. Statistical Methodology Specification

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if participants have well defined plasma profiles).

## **Endpoint / Variables**

Derived PK parameters for GSK2982772 (AUC(0-24), AUC(0-7), Cmax)

## **Model Specification**

• Dose proportionality for AUC(0-24), AUC(0-7) and Cmax following the first (morning) dose will be assessed by using a power model as described below:

$$log_e(Y_{ii}) = \mu + S_i + \beta^* log_e(D_i) + \epsilon_{ii}$$

Y<sub>ii</sub>: PK parameter (AUC(0-24), AUC(0-7), Cmax) on dose j for subject i

μ: Overall mean (intercept)

β: slope for loge transformed dose

 $S_i$ : random effect for subject i following normal distribution N(0,  $\sigma_b^2$ )

D<sub>i</sub>: dose effect (j= 60 mg, 120 mg, 240 mg)

 $\epsilon_{ij}$ : random error following normal distribution N(0,  $\sigma_w^2$ )

- The model parameters will be estimated using Restricted Maximum Likelihood with the Newton-Raphson algorithm.
- The Kenward-Roger degree of freedom approach will be used.

## **Model Checking & Diagnostics**

- If the power model has failed to converge, dose proportionality will be assessed using ANOVA.
  - Assessment of dose proportionality using ANOVA
    - The dose-normalized PK parameters (AUC(0-24), AUC(0-7), Cmax) will be calculated by dividing the PK parameters by dose.
    - The dose-normalized values will be analyzed by using the following model.

$$\log (X_{ii}) = \mu + S_i + D_i + \varepsilon_{ii}$$

 $X_{ij}$ : dose-normalized PK parameter (AUC(0-24), AUC(0-7), Cmax) on the dose i for subject i

μ : Overall mean

 $S_i$ : random effect for subject i following normal distribution N(0,  $\sigma_b^2$ )

D<sub>i</sub>: dose effect (j= 60 mg, 120 mg, 240 mg)

 $\epsilon_{ij}$  : random error following normal distribution N(0,  $\sigma_w^2)$ 

the model has dose as fixed effect and subject as random effect.

Point estimates and associated 90% confidence intervals for the differences 60 mg

 120 mg, 240 mg – 120 mg will be construced using the residual variance. These confidence intervals will then be exponentially back-transformed to provide point estimates and associated 90% confidence intervals for the ratio 60 mg/120 mg and 240 mg/120 mg.

#### **Model Results Presentation**

 The point estimates of the slope for each parameter and their 90% confidence intervals will be presented.

## 8.1.6. Details of Planned Pharmacokinetic Displays

#### Plasma Concentration-Time Data

The plasma concentrations at every scheduled time point will be summarized using n, mean, standard deviation, median, minimum, and maximum.

## Derived Plasma Pharmacokinetic Parameters (non-transformed)

The plasma pharmacokinetic parameters (AUC(0-7), AUC(7-14), AUC(14-24), AUC(0-24), Cmax, Tmax, t1/2, C0, C7, C14, C24) will be summarized using n, mean, 95% CI, standard deviation, median, minimum, and maximum.

## Derived Plasma Pharmacokinetic Parameters (log-transformed)

For each pharmacokinetic parameters with a log-normal distribution (AUC(0-7), AUC(7-14), AUC(14-24), AUC(0-24), Cmax, t1/2, C0, C7, C14, C24), the log-transformed parameters will be summarized using n, geometric mean, 95% CI of geometric mean, standard deviation of log-transformed data and between subject coefficient of variation (%CVb).

<u>Power Model Analysis for Dose Proportionality of Pharmacokinetic Parameters AUC(0-24), AUC(0-7) and Cmax</u>

The analysis results will be presented as described in Section 8.1.5.1.

## 9. APPENDICES

# 9.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the PDMP and the data handling will be determined prior to DBR.

## 9.2. Appendix 2: Schedule of Activities

## 9.2.1. Protocol Defined Schedule of Events

## Time and Events Table for Screening and Follow-up Assessments

| Procedure | Screening <sup>1</sup> | Follow-up<br>Visit <sup>2</sup> | Notes |
|---|---|---|---|
| Outpatient Visit | Х | Х | |
| Informed Consent | X | | |
| Medical/medication/drug /alcohol history | Х | | |
| Demographics | Х | | |
| Physical Examination | Х | X | Additional examinations may be performed, by the Investigators, as deemed necessary (e.g., where safety or laboratory findings indicate). |
| Drug screen | Х | | Additional tests may be performed by the Investigators, as deemed necessary (e.g., where safety or laboratory findings indicate). Tests will be conducted within site specified standards. |
| Syphilis, Human immunodeficiency virus (HIV), Human T-cell leulemia virus type 1 (HTLV-1), Hepatitis B (Hep B) and Hepatitis C (Hep C) screen | Х | | |
| Tuberculosis (TB) Test | Х | | Conducted at the standard practice of the site. |
| X-ray Test | Х | | Anterior & lateral chest X-ray will be taken. |
| Hema/Chem/Urinalysis tests | Х | Х | |
| Height and weight | Х | | |
| 12-lead ECG and vital signs | X | Х | Vital signs to include pulse rate (PR), blood pressure (BPs) and temperature. |
| AE Review | Х | Х | All Serious Adverse Effects (SAEs) will be collected from the signing of the informed consent form (ICF) until the follow-up visit at the time points specified. All AEs will be collected from the start of treatment until the follow-up visit at the time points specified. |
| Concomitant Medication Review | Х | Х | |

<sup>1:</sup> Within 30 days prior to the first dosing

<sup>2:</sup> Follow-up Visit to occur at least 7 days, and no greater than 14 days after last study treatment administration. If a participant withdrew from the study after received GSK2982772 or placebo dose, the safety assessments listed at follow-up visit will be required.

205037

# Detailed Time and Events Table for Days 1-4 (common Period1-4)

| | | | | | | | | | | | | | Day | 1 | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure <sup>1</sup> | Da<br>y<br>-1 | Pre-<br>dose | 0 | 20<br>min | 40<br>min | 1<br>hr | 1.5<br>hr | 2<br>hr | 3<br>hr | 4<br>hr | 5<br>hr | 7<br>hr | 7 hr<br>20<br>min | 7 hr<br>40<br>min | 8<br>hr | 8.5<br>hr | 9<br>hr | 10<br>hr | 12<br>hr | 14<br>hr | 14<br>hr<br>20<br>min | 14<br>hr<br>40<br>min | 15<br>hr | 15.5<br>hr |
| Admission | Χ | | | | | | | | | | | | | | | | | | | | | | | |
| Physical<br>Examination | Χ | Х | | | | | | | | | | | | | | | | | X6 | | | | | |
| Hema/Chem/<br>Urinalysis tests | Χ | | | | | | | | | | | | | | | | | | | | | | | |
| Vital signs <sup>2</sup> | | Х | | | | | | Χ | | | | | | | | | | | Х | Х | | | | |
| 12-lead ECG | | Х | | | | | | Χ | | | | | | | | | | | X5 | Х | | | | |
| Cardiac telemetry | | <=== | ==== | ===== | ===== | | ===== | ===== | | ===== | | ====== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ===== | ==== |
| PK blood sampling | | Х | | Х | Х | Х | Χ | Χ | Χ | | Х | Х | Х | Χ | Х | Х | Χ | Х | Х | Х | Х | Χ | Χ | Х |
| Neurological<br>Examination | Х | | | | | | | Х | | | | | | | | | | | | Х | | | | |
| Study<br>Treatment | | | Χ | | | | | | | | | Х | | | | | | | | Х | | | | |
| Pharmacogene tic Sample (PGx) <sup>3</sup> | | <pre>&lt;====================================</pre> | | | | | | | | | | | | | ==== | | | | | | | | | |
| Meals Served | Χ | | | | | | | | | <b>\</b> | <b>(</b> 6 | _ | _ | _ | | | | <b>\</b> | <b>(</b> 7 | | | | | |
| AE Review <sup>4</sup> | <=== | Carrier series and the series of the seri | | | | | | | | | | | | | | | | | | | | | | |
| Concomitant<br>Medication<br>Review | <=== | < | | | | | | | | | | | | | | | | | | | | | | |
| Discharge | | | | | | | | | | | | | | | | | | | | | | | | |

205037

| | | | | Da | y 2 | | | | Day | Day 4 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure 1 | 16 hr | 17 hr | 19 hr | 22 hr | 24 hr | 28 hr | 32 hr | 36 hr | 48 hr | 60 hr | 72 hr |
| Admission | | | | | | | | | | | |
| Physical Examination | | | | | Х | | | Х | Х | | Х |
| Hema/Chem/<br>Urinalysis tests | | | | | | | | | | | Х |
| Vital signs <sup>2</sup> | | | | | Х | | | | Х | | Х |
| 12-lead ECG | | | | | X | | | | X | | Х |
| Cardiac telemetry | ======== | ========= | | ======== | ======> | | | | | | |
| PK blood sampling | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Neurological<br>Examination | | | | | Х | | | | Х | | Х |
| Study Treatment | | | | | | | | | | | |
| Pharmacogenetic<br>Sample (PGx) <sup>3</sup> | ======= | | | | ======== | | ======== | ======== | -======= | | ======> |
| Meals Served | | | | | X8 | X8 | X8 | | X8 | X8 | |
| AE Review <sup>4</sup> | ======= | | | | | | | | | | ======> |
| Concomitant<br>Medication<br>Review | ======= | ======== | ======== | ======= | ======== | ======== | ======== | ========= | | | ======> |
| Discharge | | | | | | | | | | | Х |

- 1: In this study, baseline is Day -1 and Day 1 pre-dose tests.
- 2: Vital signs include PR, BPs and temperature. A 14 hr time point is to be performed prior to third dose.
- 3: A PGx blood sample will be collected at any time during the study after randomization. The participation is optional for each subject.
- 4: All SAEs will be collected from the signing of the ICF until the follow-up visit at the time points specified. All AEs will be collected from the start of treatment until the follow-up visit at the time points specified
- 5: Physical Examination and 12-lead ECG of 14hr time point are to be performed prior to third dose.
- 6: On Day 1, lunch will be served between 2 to 3 hr prior second dose.
- 7: On Day1, dinner will be served between 2 to 3 hr prior to third dose.
- 8: On Day 2-3, meal will be served per unit schedule. Mealtime will be described in SRM.

# 9.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

## 9.3.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the date of dosing date.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Previous Day of Dosing Date in Period 1 |
| Period 1 | Previous Day of Dosing Date in Period 1 ≤ Date < Previous Day of Dosing Date in Period 2 |
| Period 2 | Previous Day of Dosing Date in Period 2 ≤ Date < Previous Day of Dosing Date in Period 3 |
| Period 3 | Previous Day of Dosing Date in Period 3 ≤ Date < Previous Day of Dosing Date in Period 4 |
| Period 4 | Previous Day of Dosing Date in Period 4 ≤ Date |

## 9.3.1.1. Study Phases for Adverse Events

| Study Phase | Definition |
|---|---|
| Pre-Treatment | AE Onset Date and Time < Study First Dosing Date and Time |
| Period 1 | Dosing Date and Time in Period 1 $\leq$ AE Onset Date and Time < Dosing Date and Time in Period 2 |
| Period 2 | Dosing Date and Time in Period 2 $\leq$ AE Onset Date and Time < Dosing Date and Time in Period 3 |
| Period 3 | Dosing Date and Time in Period 3≤ AE Onset Date and Time < Dosing Date and Time in Period 4 |
| Period 4 | Dosing Date and Time in Period 4≤ AE Onset Date and Time |
| Time since Study<br>First Dose (min) | If study phase of the event is pre-treatment, AE Onset Date and Time - Study First Dosing Date and Time 1 otherwise AE Onset Date and Time – Study First Dosing Date and Time + 1 min |
| Time since Period | If study phase of the AE is pre-treatment, set to missing |
| First Dose (min) | If study phase of the AE is period 1, |
| | AE Onset Date and Time – Dosing Date and Time in Period 1 + 1 min If study phase of the AE is period 2, |
| | AE Onset Date and Time – Dosing Date and Time in Period 2 + 1 min If study phase of the AE is period 3, |
| | AE Onset Date and Time – Dosing Date and Time in Period 3 + 1 min If study phase of the AE is period 4, |
| | AE Onset Date and Time – Dosing Date and Time in Period 4 + 1 min |
| Time since Last | If study phase of the AE is pre-treatment, set to missing |
| Dose (min) | If study phase of the AE ≥ Study Last Dosing Start Date and Time, AE Onset Date and Time – Study Last Dosing Start Date and Time+ 1 min |
| Duration (min) | AE Resolution Date and Time – AE Onset Date and Time + 1 min |
| Drug-related | If relationship is marked 'YES' on eCRF or value is missing. |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be treatment emergent.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

## 9.3.1.2. Study Phases for Concomitant Medication

The study phase for concomitant medication will be categorized into pre-treatment, period 1, period 2, period 3, and period 4 based on medication start date and time.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Start Date and Time < Dosing Date in Period 1 |
| Period 1 | Dosing Date in Period 1 ≤ Start Date and Time < Dosing Date in Period 2 |
| Period 2 | Dosing Date in Period 2 ≤ Start Date and Time < Dosing Date in Period 3 |
| Period 3 | Dosing Date in Period 3 ≤ Start Date and Time < Dosing Date in Period 4 |
| Period 4 | Dosing Date in Period 4 ≤ Start Date and Time |

#### NOTES:

 Please refer to Appendix 6: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 9.4. Appendix 4: Data Display Standards & Handling Conventions

## 9.4.1. Reporting Process

| Coffeen | |
|---|---|
| Software | |
| The currently supported versions of SAS software [Insert Other Software as Required] will be used. | |
| Reporting Area | |
| HARP Server | : N/A |
| HARP Compound | : N/A |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.0.</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated | |

### 9.4.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
  - For [Insert Endpoint / Parameter] the following DP's places will be applied:
  - Summary Statistics:
  - Listings:

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

| Unscheduled Visits | |
|---|---|
| Unscheduled visi | Unscheduled visits will not be included in summary tables and/or figures. |
| All unscheduled v | All unscheduled visits will be included in listings. |
| Descriptive Summar | Descriptive Summary Statistics |
| Continuous Data | Data Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | porical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |
| <ul> <li>[Insert as Required: If any publication related displays have been specified, please provide relevant<br/>details]</li> </ul> | |

## 9.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Office function will be created according to GUI_51487. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Parameter Derivation | |
| PK Parameter to be<br>Derived by<br>Programmer | The following PK parameters will be derived by the Programmer: [C0, C7, C14, C24] |
| Pharmacokinetic Para | Pharmacokinetic Parameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to GUI_51487. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to [Insert document name] |

## 9.5. Appendix 5: Derived and Transformed Data

#### 9.5.1. **General**

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
- Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

#### **Period Day**

- Calculated as the number of days from Dosing Date in each period. For study phase derivation, see Appendix 3.
  - If Study Phase of Ref Assessment or Event = Pre-Treatment or Missing
    - $\rightarrow$  Period Day = Missing
  - If Study Phase of Ref Assessment or Event = Period X and Ref Date is on or after Dosing Date in Period X
    - → Period Day = Ref Date Dosing Date in Period X + 1 day
  - If Study Phase of Ref Assessment or Event = Period X and Ref Date is before Dosing Date in Period X
    - $\rightarrow$  Period Day = Ref Date Dosing Date in Period X

Note: X takes a value of 1, 2, 3, 4.

## 9.5.2. Study Population

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - o A date and month will be imputed as '30th June' as it will not be captured.
- Date of Informed Consent will be used as reference date of calculation.

## 9.5.3. Safety

#### **Laboratory Parameters**

#### **Imputation**

• If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.

o Example 1: 2 Significant Digits = '< x' becomes x - 0.01o Example 2: 1 Significant Digit = '> x' becomes x + 0.1o Example 3: 0 Significant Digits = '< x' becomes x - 1

 The default convention for reporting of clinical laboratory units will be the international system of units (SI units).

## 9.6. Appendix 6: Reporting Standards for Missing Data

## 9.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as completion of all phases of the study including the last visit or the last scheduled procedure.</li> <li>Withdrawn subjects may be replaced in the study.</li> </ul> |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |

## 9.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 9.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing.</li> <li>The eCRF allows for the possibility of missing times to be recorded for AE start and end dates. Missing dates will be imputed using the following convention: <ul> <li>If the missing time is a start date, a '00:00' will be used for the time.</li> <li>If the missing date is a stop date, a '23:59' will be used for the time.</li> </ul> </li> <li>The recorded missing time will be displayed in listings without imputed values.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The eCRF allows for the possibility of missing times to be recorded for concomitant medications start and end dates. Missing dates will be imputed using the following convention: <ul> <li>If the missing time is a start date, a '00:00' will be used for the time.</li> </ul> </li> </ul> |

| Element | Reporting Detail |
|---|---|
| | <ul> <li>If the missing date is a stop date, a '23:59' will be used for the time.</li> </ul> |
| | The recorded partial date and missing time will be displayed in listings without imputed values. |

# 9.7. Appendix 7: Values of Potential Clinical Importance

## 9.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Hometoorit | Ratio of | | | 0.54 |
| Hematocrit | 1 | $\Delta$ from BL | ↓ 0.075 | |
| Lloomodobin | g/L | | | 180 |
| Haemoglobin | | $\Delta$ from BL | ↓ 25 | |
| Lymphocytes | x109/ L | | 0.8 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| White Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |
## 9.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | Absolute | | |
| Absolute QTc Interval | msec | | > 450 [1] |
| Absolute PR Interval | msec | < 110 [1] | > 220 [1] |
| Absolute QRS Interval | msec | < 75 [1] | > 110 [1] |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | > 60 [1] |

## NOTES:

## 9.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

<sup>1.</sup> Represent standard ECG values of PCI for HV studies

# 9.8. Appendix 8: Abbreviations & Trade Marks

## 9.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| ITT | Intent-To-Treat |
| PCI | Potential Clinical Importance |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| TFL | Tables, Figures & Listings |

## 9.8.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin |

## 9.9. Appendix 9: List of Data Displays

## 9.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|------------|
| Study Population | 1.1 to 1.7 | - |
| Safety | 2.1 to 2.21 | - |
| Pharmacokinetic | 3.1 to 3.5 | 3.1 to 3.5 |
| Section | Listings | |
| ICH Listings | 1 to 37 | |

## 9.9.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 10: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|-----------------|--------|--------|---------|
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Safety | SAF_Fn | SAF_Tn | SAF_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 9.9.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

205037

# 9.9.4. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | • |
| 1.1. | Safety | ES1A | Summary of Subject Disposition for the Participant Conclusion Record | ICH E3, FDAAA, EudraCT | SAC |
| 1.2. | Enrolled | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC |
| 1.3. | Enrolled | NS1 | Summary of Number of Participant by Country and Site ID | EudraCT/Clinical Operations | SAC |
| Protoc | ol Deviation | | | | • |
| 1.4. | Safety | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| Demog | Demographic and Baseline Characteristics | | | | |
| 1.5. | Safety | DM3 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC |
| 1.6. | Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC |
| 1.7. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | SAC |

205037

# 9.9.5. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 2.1. | Safety | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| 2.2. | Safety | AE5A | Summary of All Adverse Events by Maximum Intensity by System Organ Class and Preferred Term | ICH E3 | SAC |
| 2.3. | Safety | AE1CP | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| 2.4. | Safety | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | ICH E3 | SAC |
| Labora | tory: Chemistry | <i>y</i> | | | |
| 2.5. | Safety | LB1 | Summary of Chemistry Values | | SAC |
| 2.6. | Safety | LB1 | Summary of Chemistry Changes from Baseline | ICH E3 | SAC |
| 2.7. | Safety | LB4 | Summary of Chemistry Data Shifts from Baseline Relative to PCI Criteria | ICH E3 | SAC |
| Labora | tory: Hematolo | gy | | | |
| 2.8. | Safety | LB1 | Summary of Hematology Values | | SAC |
| 2.9. | Safety | LB1 | Summary of Hematology Changes from Baseline | ICH E3 | SAC |
| 2.10. | Safety | LB4 | Summary of Hematology Data Shifts from Baseline Relative to PCI Criteria | ICH E3 | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Urinalysis | 3 | | | |
| 2.11. | Safety | LB1 | Summary of Urinalysis Data (Gravity and pH) | | SAC |
| 2.12. | Safety | LB1 | Summary of Urinalysis Concentration Change from Baseline (Gravity and pH) | ICH E3 | SAC |
| 2.13. | Safety | UR3b | Summary of Urinalysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, Urobilinogen) | | SAC |
| Neurol | ogical Examina | tion | | | <u> </u> |
| 2.14. | Safety | NE1 | Summary of Neurological Examination | | SAC |
| ECG | | | | | · |
| 2.15. | Safety | EG1 | Summary of ECG Findings | IDSL | SAC |
| 2.16. | Safety | EG2 | Summary of ECG Values | | SAC |
| 2.17. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | SAC |
| 2.18. | Safety | HM1 | Summary of Cardiac Telemetry | IDSL | SAC |
| 2.19. | Safety | HM2 | Summary of Cardiac Telemetry Abnpormalities | IDSL | SAC |
| Vital Si | gns | | | | |
| 2.20. | Safety | VS1 | Summary of Vital Signs | IDSL | SAC |
| 2.21. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | SAC |

205037

## 9.9.6. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.1. | PK | PK01 | Summary of GSK2982772 Plasma Pharmacokinetic Concentration-Time Data | | SAC |
| 3.2. | PK | PK03 | Summary of Derived GSK2982772 Pharmacokinetic Parameters (non-transformed) | | SAC |
| 3.3. | PK | PK05 | Summary of GSK2982772 Pharmacokinetic Parameters (log-transformed) | | SAC |
| 3.4. | PK | PK_T1 | Power Model Analysis for GSK2982772 Dose Proportionality of Pharmacokinetic Parameters (AUC(0-24), AUC(0-7), Cmax) | | SAC |
| 3.5. | PK | PK_T2 | ANOVA Model Analysis for GSK2982772 Dose Proportionality of Dose-Normalized Derived Pharmacokinetic Parameters(AUC(0-24), AUC(0-7), Cmax) | This table will be provided if the power model fails to converge. | SAC |

205037

## 9.9.7. Pharmacokinetic Figures

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.1. | PK | PK16b | Individual GSK2982772 Plasma Concentration–Time Plots by Subject | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 3.2. | PK | PK24 | Individual GSK2982772 Plasma Concentration–Time Plots by Treatment | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 3.3. | PK | PK17 | Mean (+SD) GSK2982772 Plasma Concentration–Time Plots | A graph on linear and semi-logarithmic scales will be produced. SD will also be displayed. | SAC |
| 3.4. | PK | PK18 | Median GSK2982772 Plasma Concentration–Time Plots | A graph on linear and semi-logarithmic scales will be produced. | SAC |
| 3.5. | PK | PK28 | Plot of Individual (+Geometric Mean and 95% CIs) GSK2982772<br>Pharmacokinetic Parameters (AUC(0-24), AUC(0-7), Cmax)<br>versus Dose | | SAC |

205037

# 9.9.8. ICH Listings

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | Safety | ES3 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 3. | Safety | SD3 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC |
| 4. | Safety | BL2 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | SAC |
| 5. | Safety | TA2 | Listing of Planned and Actual Treatments | IDSL | SAC |
| Protoc | ol Deviations | | | 1 | |
| 6. | Safety | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 7. | Safety | IE4 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Popula | tions Analysed | | | | |
| 8. | Safety | SP3A | Listing of Subjects Excluded from Any Population | ICH E3 | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 9. | Safety | DM4 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 10. | Safety | DM10 | Listing of Race | ICH E3 | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 11. | Safety | MH3 | Listing of Medical Conditions | IDSL | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 12. | Safety | CM5 | Listing of Concomitant Medications | IDSL | SAC |
| Exposu | re and Treatmo | ent Compliance | | | |
| 13. | Safety | EX4 | Listing of Exposure Data | ICH E3 | SAC |
| Advers | e Events | | | | |
| 14. | Safety | AE9CP | Listing of All Adverse Events | ICH E3 | SAC |
| 15. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |
| 16. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| Serious | s and Other Sig | nificant Adverse | -<br>Events | | |
| 17. | Safety | AE9CP | Listing of Fatal Serious Adverse Events | ICH E3 | SAC |
| 18. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC |
| Hepato | biliary (Liver) | | | , | |
| 19. | Safety | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | SAC |
| 20. | Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | SAC |
| Chemis | stry | 1 | | | 1 |
| 21. | Safety | LB6 | Listing of All Chemistry Data | ICH E3 | SAC |
| 22. | Safety | LB6 | Listing of All Chemistry Data for Subjects with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| 23. | Safety | LB6 | Listing of Chemistry Values of Potential Clinical Importance | | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Haema | tology | | | | |
| 24. | Safety | LB6 | Listing of All Haematology Data | ICH E3 | SAC |
| 25. | Safety | LB6 | Listing of All Haematology Data for Subjects with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| 26. | Safety | LB6 | Listing of Haematology Values of Potential Clinical Importance | | SAC |
| Urinary | /sis | | | | |
| 27. | Safety | LB6 | Listing of Urinarysis Data (Gravity and pH) | | SAC |
| 28. | Safety | LB14 | Listing of Urinarysis Data (Glucose, Protein, Blood, Ketones, Bilirubin, and Urobilinogen) | | SAC |
| Neurol | ogical Examina | tion | | | |
| 29. | Safety | NE2 | Listing of Neurological Examinations | IDSL | SAC |
| ECG | | | | | |
| 30. | Safety | EG6 | Listing of ECG Findings | | SAC |
| 31. | Safety | EG4 | Listing of All ECG Values | IDSL | SAC |
| 32. | Safety | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | IDSL | SAC |
| 33. | Safety | HM10 | Listing of Clinically Significant Cardiac Telemetry Abnormalities | IDSL | SAC |
| Vital Si | gns | | | | |
| 34. | Safety | VS5 | Listing of All Vital Signs Data | IDSL | SAC |
| 35. | Safety | VS5 | Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance | IDSL | SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharmacokinetics | | | | | |
| 36. | PK | PK08 | Listing of GSK2982772 Plasma Pharmacokinetic Concentration-<br>Time Data | IDSL | SAC |
| 37. | PK | PK14 | Listing of Derived GSK2982772 Plasma Pharmacokinetic Parameters | IDSL All PK parameters in Section 8.1.1.2 will be provided in a listing | SAC |

205037

## 9.10. Appendix 10: Example Mock Shells for Data Displays

Example: PK\_T1
Protocol: 205037

Page 1 of 1

Protocol: 20503 Population: PK

Table x.x

Power Model Analysis for GSK2982772 Dose Proportionality of Pharmacokinetic Parameters (AUC(0-24), AUC(0-7), Cmax)

| Parameter | Effect | n<br>I | Slope<br>Point Estimate | 90% CI |
|------------|------------------|--------|-------------------------|----------|
| AUC (0-24) | Log(dose levels) | XX | XXX | (xx,xx) |
| AUC(0-7) | Log(dose levels) | XX | XXX | (xx, xx) |
| Cmax | Log(dose levels) | XX | xxx | (xx, xx) |

Note: The power model was fitted to loge-transformed PK parameters with loge-transformed dose as fixed effet. The slope with corresponding 90% confidence interval was estimated from the power model to assess the degree of dose-proportionality (slope around unity indicates dose-proportionality).

PPD

205037

Example: PK\_T2
Protocol: 205037

Protocol: 205037 Page 1 of 1 Population: PK

Table x.x

ANOVA Model Analysis for GSK2982772 Dose Proportionality of Dose-Normalized Derived Pharmacokinetic Parameters (AUC(0-24), AUC(0-7), Cmax)

| Parameter | Treatment Comparison | Ratio of<br>Adjusted Geo.<br>Means | 90% CI |
|---|---|---|---|
| AUC (0-24) | 60 mg / 120 mg | X.XXX | (x.xxx,x.xxx) |
| | 240 mg / 120 mg | x.xxx | (x.xxx,x.xxx) |
| AUC (0-7) | 60 mg / 120 mg | x.xxx | (x.xxx,x.xxx) |
| | 240 mg / 120 mg | x.xxx | (x.xxx,x.xxx) |
| Cmax | 60 mg / 120 mg | x.xxx | (x.xxx,x.xxx) |
| | 240 mg / 120 mg | X.XXX | (x.xxx,x.xxx) |

Note: The ANOVA model was fitted to loge-transformed and dose-normalized PK parameters with dose as fixed effet. The ratios of adjusted geographic means with corresponding 90% confidence interval were estimated from the ANOVA model to assess the degree of dose-proportionality (slope around unity indicates dose-proportionality).

PPD